CLINICAL TRIAL: NCT00133367
Title: Phase II Study of Sequential Unrelated Cord Blood Transplantation Using Tacrolimus and Sirolimus as Graft Versus Host Disease Prophylaxis
Brief Title: Study of Unrelated Cord Blood Transplantation Using Tacrolimus and Sirolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Karen Ballen, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-154
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Myeloma; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Myelogenous Leukemia; Lymphoblastic Leukemia
Keywords: Hematologic malignancy; Cord blood transfusion; Graft versus host disease; tacrolimus; sirolimus
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Myeloid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms; Graft vs Host Disease | interventions — Tacrolimus; Sirolimus; Granulocyte Colony-Stimulating Factor; Antilymphocyte Serum; thymoglobulin; fludarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tacrolimus — Given three days before transplant and every day for 3-6 months after transplant. After first 100 days post-transplant, the dose will be reduced.
Drug: Sirolimus — Given three days before transplant and every day for 3-6 months after transplant. After first 100 days post-transplant, the dose will be reduced.
Drug: G-CSF — Given starting on day 5 after transplant until the subjects white blood cell count recovers.
Drug: Antithymocyte globulin — Given intravenously for 4 days before transplant (days 7, 5, 3, 1).
Drug: Thymoglobulin — Given intravenously for 4 days before transplant (days 7, 5, 3, 1).
Drug: Fludarabine — Given intravenously for six days prior to transplant (days 8,7,6,5,4,3).
Drug: Melphalan — Given intravenously on day 2 before transplant.

SUMMARY:
The purpose of this study is to measure the effectiveness of 2 drugs, tacrolimus and sirolimus, in preventing graft versus host disease (GVHD) after treatment with chemotherapy followed by donor cord blood transplantation.

DETAILED DESCRIPTION:
* The chemotherapy portion of the study involves the intravenous administration of fludarabine, for six days (Days 8, 7, 6, 5,4, and 3) before transplant, melphalan, for one day (Day 2) before transplant. Antithymocyte globulin, or thymoglobulin, will be given IV daily for 4 days (days 7, 5, 3, and 1 before transplant). This drug also helps to suppress the immune system, allowing the cord blood cells to grow and reproduce.
* Immunosuppression therapy consists of the drugs tacrolimus and sirolimus. The patient will receive these 3 days before the transplant and every day for 3-6 months after transplant. After the first 100 days post transplant, the doses of tacrolimus and sirolimus will begin to be reduced with the goal of having the patient off both drugs by 6-9 months after transplant.
* After completion of conditioning therapy described above, the patient will receive 2 cord blood units 1-6 hours apart. To help with engraftment, the patient will also receive G-CSF starting on day five after transplant, until the patients white blood cells recover.
* Follow-up visits will continue every 6 months after the last treatment dose and will last up to 2 years.
* Blood tests will be drawn frequently to test whether the donor's immune cells have engrafted as well as to test the levels of Tacrolimus and Sirolimus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies for whom allogeneic stem cell transplantation is deemed clinically appropriate
* Non-Hodgkin's lymphoma, or Hodgkin's lymphoma: in Complete Remission >2 (second complete remission, third complete remission, etc) or in partial remission
* Multiple myeloma: relapsed
* Chronic lymphocytic leukemia, Rai stage III or IV, or lymphocyte doubling time of 6 months, or stage I-II, having progressed after > 2 chemotherapy regimens, in partial remission.
* Acute myelogenous or lymphoblastic leukemia in second or subsequent remission or in first remission with adverse cytogenetic or antecedent hematologic disorder
* Chronic myelogenous leukemia in accelerated or second stable phase, or imatinib resistant and not eligible for an ablative transplant
* Myelodysplasia, previously treated or not eligible for ablative transplant
* Age 18-65 years.
* ECOG performance status of 0, 1, or 2.
* Lack of 6/6 or 5/6 HLA-matched related, 10/10 matched unrelated donor, or unrelated donor not available within the time frame necessary to perform a potentially curative stem cell transplant.

Exclusion Criteria:

* Cardiac disease:

  * symptomatic congestive heart failure or
  * radionuclide ventriculogram (RVG) or echocardiogram determined left ventricular ejection fraction of < 40%,
  * active angina pectoris, or
  * uncontrolled hypertension.
* Pulmonary disease:

  * severe chronic obstructive lung disease, or
  * symptomatic restrictive lung disease, or
  * corrected DLCO of < 50% of predicted.
* Renal disease:

  * serum creatinine > 2.0 mg/dl.
* Hepatic disease:

  * serum bilirubin > 2.0 mg/dl (except in the case of Gilbert's syndrome or hemolytic anemia in which the bilirubin can be elevated greater than 2.0mg/dl),
  * SGOT or SGPT > 3 x normal.
* Neurologic disease:

  * symptomatic leukoencephalopathy,
  * active central nervous system (CNS) malignancy or other neuropsychiatric abnormalities believed to preclude transplantation (previous CNS malignancy, presently in complete remission [CR] is not exclusion).
* HIV antibody.
* Uncontrolled infection.
* Pregnancy or breast feeding mother.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of tacrolimus and sirolimus in preventing graft versus host disease | 2 years

SECONDARY OUTCOMES:
To evaluate the days to neutrophil engraftment and platelet engraftment | 2 years
To evaluate the relapse rate and overall disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Ballen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Brown JA, Stevenson K, Kim HT, Cutler C, Ballen K, McDonough S, Reynolds C, Herrera M, Liney D, Ho V, Kao G, Armand P, Koreth J, Alyea E, McAfee S, Attar E, Dey B, Spitzer T, Soiffer R, Ritz J, Antin JH, Boussiotis VA. Clearance of CMV viremia and survival after double umbilical cord blood transplantation in adults depends on reconstitution of thymopoiesis. Blood. 2010 May 20;115(20):4111-9. doi: 10.1182/blood-2009-09-244145. Epub 2010 Jan 27. PMID 20107229